CLINICAL TRIAL: NCT00000771
Title: A Double-Blind, Placebo-Controlled Trial of Paromomycin for Treatment of Cryptosporidiosis in Patients With Advanced HIV Disease and CD4 Counts Under 150 Cells/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 192; 11167 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: Cryptosporidiosis; Acquired Immunodeficiency Syndrome; Paromomycin
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Paromomycin

INTERVENTIONS:
Drug: Paromomycin sulfate

SUMMARY:
To determine the effectiveness of oral paromomycin sulfate for 21 days compared to placebo in the treatment of cryptosporidiosis in patients with HIV infection. To evaluate the safety of oral paromomycin at two different doses. To explore whether paromomycin administered over a longer period provides additional benefit.

In previous studies, patients with cryptosporidiosis demonstrated dramatic improvement with paromomycin therapy.

DETAILED DESCRIPTION:
In previous studies, patients with cryptosporidiosis demonstrated dramatic improvement with paromomycin therapy.

Patients are randomized to receive either placebo or paromomycin for 3 weeks. After the initial double-blind phase, all patients receive open-label paromomycin for 3 weeks. Following 6 weeks of therapy, patients who do not achieve a complete response receive a higher dose of paromomycin for an additional 3 weeks, while complete responders continue receiving the original dose for an additional 3 weeks. Complete or partial responders after 9 weeks may receive 16 additional weeks of optional maintenance therapy at the dose at which their response was achieved. Treatment continues for up to 25 weeks total. Patients are followed at weeks 1, 3, 4, 6, 7, and 9, and then at 2-4 week intervals.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Macrolides for disseminated Mycobacterium avium.
* Atovaquone for toxoplasmosis.
* Other antimicrobials for concurrent infections.
* Lomotil, Imodium, or deodorized opium tincture in a standardized regimen for diarrhea.

Patients must have:

* Advanced HIV disease.
* Diarrhea presumptively caused by Cryptosporidia.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Hypersensitivity to aminoglycosides.
* Inability to swallow capsules.
* Active infection due to other enteric pathogens. Previous diagnosis of CMV or MAC infection permitted if patient is currently stabilized on a therapeutic regimen (clarithromycin up to 500 mg bid or azithromycin up to 600 mg daily).
* Other known causes for diarrhea (e.g., malabsorption syndrome, gastrointestinal Kaposi's sarcoma).

Concurrent Medication:

Excluded during the first 9 weeks of study:

* Agents with putative anticryptosporidial activity (such as spiramycin, diclazuril, letrazuril, or bovine colostrum).
* Octreotide acetate (Sandostatin).
* Antidiarrheals other than those specifically allowed.
* Clarithromycin if initiated at 500 mg or higher or azithromycin if initiated at 600 mg or higher.

Prior Medication:

Excluded:

* Paromomycin at > 1 g/day for >= 14 days prior to study entry.

Excluded within 14 days prior to study entry:

* Agents with putative anticryptosporidial activity (such as spiramycin, diclazuril, letrazuril, or bovine colostrum), with the exception of macrolides that are permitted for other indications.
* Octreotide acetate (Sandostatin).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68
Dates: Study Completion 1996-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey J, Study Chair
Locations (15):
- United States (14):
  - USC CRS, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Weiss Memorial Hosp., Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Washington U CRS, St Louis, Missouri
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Hewitt RG, Yiannoutsos CT, Higgs ES, Carey JT, Geiseler PJ, Soave R, Rosenberg R, Vazquez GJ, Wheat LJ, Fass RJ, Antoninievic Z, Walawander AL, Flanigan TP, Bender JF. Paromomycin: no more effective than placebo for treatment of cryptosporidiosis in patients with advanced human immunodeficiency virus infection. AIDS Clinical Trial Group. Clin Infect Dis. 2000 Oct;31(4):1084-92. doi: 10.1086/318155. Epub 2000 Oct 25. PMID 11049793